CLINICAL TRIAL: NCT01270620
Title: Desflurane or Propofol Anesthesia in Elderly Obese Patients Undergoing Total Knee Replacement: A Pilot Assessment of Short-term and Long-term Differences in Outcome
Brief Title: Desflurane or Propofol Anesthesia in Elderly Obese Patients Undergoing Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pedro Paulo Tanaka (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pedro Paulo Tanaka, Clinical Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SU-12062010-7277; IRB: 4593 (Other: Stanford Instituinal Review Board); SPO: 48391 (Other: Sponsored Project Office Stanford University)
Record Dates: First submitted 2010-12-14; First posted 2011-01-05 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Arthritis
Keywords: elderly obese
MeSH Terms: conditions — Obesity; Arthritis | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Patients will receive propofol as general anesthetics.
  Interventions: Drug: propofol
- Desflurane (Active Comparator): Patients will receive desflurane as general anesthetics.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: propofol — comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
  Arms: Propofol
Drug: Desflurane — comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
  Other Names: Suprane
  Arms: Desflurane

SUMMARY:
You are invited to participate in a research study assessing your mental status in the first days after your surgery and how you will be doing in the 2 years following the surgery. The investigators hope to learn more about the incidence of postoperative confusion and a possible relation with 2 anesthesia techniques that are routinely used. The first one is an anesthesia technique that uses the inhaled anesthetic gas desflurane and the second one is an anesthesia technique that uses the anesthetic propofol administered by infusion in a vein. The investigators are also looking to see if there is a relationship between anesthesia technique and cardiovascular outcomes. You were selected as a possible participant in this study because at your age this phenomenon appears to have a greater incidence.

DETAILED DESCRIPTION:
Trial Objectives:

This will be a randomized, prospective, single-center, assessor blinded pilot study comparing two different anesthesia techniques in 100 elderly obese patients undergoing primary total knee arthroplasty.

Endpoints:

* The incidence of postoperative delirium as measured by the Confusion Assessment Score. Confusion assessment score will be administered at baseline, one hour after arrival in the post anesthesia care unit and 6-8, 24 and 48 hrs postoperatively.
* Cognitive function as measured by Test for Attentional Performance, Digit-Symbol-Substitution Test, Recal of Digit Span , Well-being Test BF-S, Spielberger State-Trait Anxiety Inventory and the Trail Making Test A and B. Cognitive function tests will be administered at baseline, 6-8 and 48 hrs post operatively. Postoperative Cognitive Dysfunction is defined as a 20% decline of the baseline values.

Intraoperative

* Sensory block (femoral)
* Blood pressure
* Heart rate
* Patient state index values
* Degree of neuromuscular blockade
* Esophageal temperature
* End tidal concentration of CO2
* End tidal concentration of desflurane
* Amount of vasopressors (ephedrine or phenylephrine)
* Amount of intravascular fluid administration
* Dose and mean infusion rates of all IV drugs (propofol)
* Duration of anesthesia
* Duration of surgery
* Time to spontaneous breathing after desflurane/propofol discontinuation
* Time to eye opening after desflurane/propofol discontinuation
* Time to tracheal extubation after desflurane/propofol discontinuation
* Time to following command after desflurane/propofol discontinuation

Post operative

* Nausea and vomiting: one hour after arrival in the post anesthesia care unit and 6-8, 24 and 48 hrs postoperatively
* Pain visual analogue score measured one hour after arrival in the post anesthesia care unit and 6-8, 24 and 48 hrs postoperatively
* Recovery room time
* Amount of local anesthetics (ropivacaine)
* Amount of opioids (Patient controlled analgesia hydromorphone)

Cardiovascular

* B-type natriuretic peptide measured preoperatively and on postoperative days 1 and 2
* N-terminal proB-type natriuretic peptide measured preoperatively and on postoperative days 1 and 2
* Troponin I measured preoperatively and on postoperative days 1 and 2
* Patients will be followed by a blinded investigator for a 2 year period to record the development of cardiac complications defined by a broad composite that included cardiac death and nonfatal myocardial infarction. Cardiac composite including: all-cause mortality, acute myocardial infarction, unstable angina, congestive heart failure, new atrial or ventricular dysrhythmia requiring treatment, and cerebrovascular insult.

Protocol This will be a randomized, prospective, single-center, assessor blinded study comparing two different anesthesia techniques in 100 elderly obese patients undergoing primary total knee arthroplasty. We expect to enroll all patients in a 2 year period.

The study will be performed according to the Declaration of Helsinki principles, and written informed consent will be obtained from each patient. Preoperatively baseline values will be obtained for the cardiovascular, mental status, respiratory and pain outcome measures.

Mental status: During their preoperative visit patients will be given the neuropsychological tests in the following order: 1. Confusion Assessment Method . The confusion assessment method is a screening instrument for delirium consisting of four clinical criteria: (1) acute onset and fluctuating course, (2) inattention, (3) disorganized thinking, and (4) altered level of consciousness. For a person to be considered delirious, both the first and the second criteria and either the third or the fourth criteria have to be present. The confusion assessment method has a high inter-observer reliability (0.8 -1.0), a sensitivity of 94-100%, and a specificity of 90-95%. 2. Modified Mini-Mental State Examination. This extended measure of general cognition was developed to overcome shortcomings of the traditional Mini-Mental State Examination score, specifically its ceiling effects and narrow range of possible scores. The Modified Mini-Mental State Examination will be administered at the preoperative visit to assess the baseline cognitive function of the patient. 3. Computerized Test for Attentional Performance , Digit-Symbol-Substitution Test, Recall of Digit Span, Well-being Test BF-S, Spielberger State-Trait Anxiety Inventory and the Trail Making Test A and B.

Patients will be visited for the first 2 days after surgery or until discharge, whichever came first, and the confusion assessment method will be administered one hour after arrival in the post anesthesia care unit and 6-8, 24 and 48 hrs postoperatively to determine whether the patient is experiencing delirium. Each patient will be interviewed by the same trained research assistant before surgery and during the postoperative visits. We will define the occurrence of delirium as the patient meeting the confusion assessment method criteria for delirium on any of the postoperative assessments. If a patient is positive for delirium, a second member of the research team will be consulted to verify the diagnosis. Cognitive function tests will be administered, 6-8 and 48 hrs post operatively. Postoperative Cognitive Dysfunction is defined as a 20% decline of the baseline values.

Cardiovascular: Preoperative testing will include 12-lead ECG. Blood samples for Natriuretic peptide levels and N-terminal proB-type natriuretic peptide and Troponin I will be obtained at the time of the admission and on postoperative day 1 and day 2. Plasma NT-proB-type natriuretic peptide will be determined using the Elecsys proB-type natriuretic peptide sandwich immunoassay on an Elecsys 2010 (Roche Diagnostics, Basel, Switzerland). Two cut offs for NT-proB-type natriuretic peptide will be selected before the analyses, 300 pg/ml and 600 pg/ml, with a value of less than 300 pg/ml shown to be optimal for ruling out heart failure as a predictor. B-type natriuretic peptide will be determined using immunoradiometric assay kit. Values of B-type natriuretic peptide (pg/mL) 31.0 ± 2.4 are considered normal for patients over 65 years old.

After discharge from the hospital patients will be followed blindly for a 2 year period to record the development of cardiac complications defined by a broad composite that included cardiac death and nonfatal myocardial infarction. Cardiac composite including: all-cause mortality, acute myocardial infarction, unstable angina, congestive heart failure, new atrial or ventricular dysrhythmia requiring treatment, and cerebrovascular insult. Information will be collected at 1, 3, 6, 12, 18 and 24 months after surgery.

Outcome measures and postoperative complications including nausea and vomiting will be recorded by an assessor blinded to the treatment allocation.

Patients will be randomly allocated to one of two treatment groups on the day of surgery using a computer generated assignment. Group D will receive desflurane and group P will receive propofol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years old
* Body mass index > 30 kg/m2
* Undergoing primary total knee arthroplasty surgery
* American society of anesthesiology classification II-III

Exclusion Criteria:

* Patient refusal to participate in the study
* Patient refusal or failure of regional block
* Patients with preexisting neuro-cognitive disorders
* Known intolerance to any of the drugs to be used according to the study protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrikus Lemmens, Principal Investigator — Stanford University; Pedro Paulo Tanaka, Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred patients provided consented to participate in the study during June 2010 to August 2014.
Groups:
- Desflurane Group: Patients will receive desflurane as general anesthetic. Desflurane is inhaled agent which will be provided continuously via ETT in concentrations varying from 4-6% according to BIS monitoring.
  Desflurane: comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
- Propofol Group: Patients will receive propofol as general anesthetic Propofol is an intravenous agent which will be provided continuously via IV in doses varying from 100 to 200 mcg/kg/min according to BIS monitoring.
  Propofol: comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
Period: Overall Study
Arm/Group | Desflurane Group | Propofol Group
Started | 50 | 50
Completed | 49 | 47
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Desflurane; Propofol: Patients received propofol or desflurane as general anesthetic for total knee replacement.
  Inclusion criteria: Age > 65 years old; BMI > 30 kg/m2; undergoing primary total knee replacement surgery; and ASA classification II-III
- Total: Total of all reporting groups
Arm/Group | Desflurane | Propofol | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (4.0) | 71 (5.8) | 70.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 34 | 55
  Male | 29 | 16 | 45
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Delirium
Description: The primary end point was the incidence of postoperative delirium as measured by the Confusion Assessment Method (CAM).
Time Frame: 48 hours
Measure: Number; unit: participants
Groups:
- Desflurane: Patients received desflurane as general anesthetic
  propofol or desflurane: comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
- Propofol: Patients received propofol as general anesthetic
  propofol or desflurane: comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 0 | 0

2. Secondary Outcome: - Time to Spontaneous Breathing After Desflurane/Propofol Discontinuation
Time Frame: first day
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Desflurane: Patients received desflurane as general anesthetic
- Propofol: Patients received propofol as general anesthetic
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
seconds | 270 [120 to 480] | 300 [120 to 465]

3. Secondary Outcome: - Time to Eye Opening After Desflurane/Propofol Discontinuation
Time Frame: first day
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
seconds | 420 [240 to 600] | 395 [180 to 655]

4. Secondary Outcome: - Time to Tracheal Extubation After Desflurane/Propofol Discontinuation
Time Frame: first day
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Desflurane: Patient received desflurane as a general anesthesia
- Propofol: Patient received propofol as a general anesthesia
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
seconds | 420 [300 to 600] | 526 [300 to 720]

5. Secondary Outcome: - Time to Following Command After Desflurane/Propofol Discontinuation
Time Frame: first day
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
seconds | 480 [300 to 600] | 450 [240 to 660]

6. Secondary Outcome: Nausea and Vomiting
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 3 | 4

7. Secondary Outcome: Recovery Room Time
Time Frame: first day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
minutes | 65 [46 to 76] | 60.5 [45 to 83.75]

8. Secondary Outcome: B-type Natriuretic Peptide
Time Frame: Change from Baseline to day one
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
ng/L | 47 [31 to 76] | 43 [14.5 to 77.5]

9. Secondary Outcome: N-terminal proBNP
Time Frame: Change from baseline to day one
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
ng/L | 83 [46 to 159] | 86 [9 to 194]

10. Secondary Outcome: Troponin I
Description: Patients who had troponin level > 0.2 ng/mL
Time Frame: 2 days
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 1 | 0

11. Secondary Outcome: BNP
Time Frame: Change form baseline to post-operative day 2
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
ng/L | 83.5 [35.5 to 174] | 92 [45.5 to 196.5]

12. Secondary Outcome: ProBNP
Time Frame: Change from baseline to post-operative day 2
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
ng/L | 330 [147 to 682.5] | 311.5 [153.8 to 573.2]

13. Primary Outcome: Recall of Digit Span
Description: • The Digit Span subtest of the Wechsler Adult Intelligence Scale-Revised is a test that requires subjects to repeat a series of digits that have been verbally presented to them both forward and, in a later independent test, reverse order. It measures attention and working memory
Time Frame: Change > 20% from baseline to 6-8 hours after surgery
Measure: Number; unit: participants
Groups:
- Desflurane: Patients received desflurane as a general anesthetic
- Propofol: Patients received propofol as a general anesthetic
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 11 | 8

14. Primary Outcome: Recall of Digit Span
Description: as for outcome 13
Time Frame: Change > 20% from baseline to 48 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 10 | 9

15. Primary Outcome: Digit Symbol Substitution Test
Description: • The Digit Symbol Substitution Test (DSST) measures attention, working memory, sustained visual attention and psychomotor speed. Subjects are given a table that pairs digits and symbols, and asked to decipher a code using the table, completing as many as possible in 90 seconds. The DSST has been found to be more sensitive than other tests to changes in high-levels of cognition
Time Frame: Change > 20% from baseline to 6-8 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 22 | 17

16. Primary Outcome: Digit Symbol Substitution Test
Description: as for outcome 15
Time Frame: Change > 20% from baseline to 48 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 24 | 16

17. Primary Outcome: Trail Making Part A
Description: • Trail Making Test is an executive measure of sequencing and cognitive flexibility. Trail A requires the subject to rapidly sequence a straightforward series. The scoring for this test is the time in seconds required for completion of the test
Time Frame: Change > 20% from baseline to 6-8 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 25 | 25

18. Primary Outcome: Trail Making Part A
Description: as for outcome 17
Time Frame: Change > 20% from baseline to 48 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 26 | 19

19. Primary Outcome: Trail Making Part B
Description: • Trail Making Test is an executive measure of sequencing and cognitive flexibility. Trail B is a more difficult cognitive flexibility task requiring the subject to follow a sequential pattern while shifting cognitive sets and reflects executive functioning, although other cognitive abilities, such as psychomotor speed and visual scanning, are necessary for successful completion of the task. The scoring for this test is the time in seconds required for completion of the test
Time Frame: Change > 20% from baseline to 6-8 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 29 | 22

20. Primary Outcome: Trail Making Part B
Description: Trail Making Test is an executive measure of sequencing and cognitive flexibility. Trail B is a more difficult cognitive flexibility task requiring the subject to follow a sequential pattern while shifting cognitive sets and reflects executive functioning, although other cognitive abilities, such as psychomotor speed and visual scanning, are necessary for successful completion of the task. The scoring for this test is the time in seconds required for completion of the test
Time Frame: Change > 20% from baseline to 48 hours after surgery
Measure: Number; unit: participants
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
participants | 29 | 22

21. Secondary Outcome: Duration of Surgery
Time Frame: Time from Incision to closure of surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
minutes | 103.5 [91.5 to 117] | 95 [84.25 to 123]

22. Secondary Outcome: Duration of Anesthesia
Time Frame: Time from induction to extubation
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
minutes | 137.5 [121.2 to 156.5] | 133.5 [115 to 159.2]

23. Secondary Outcome: Amount of Intraoperative Fentanyl
Time Frame: From the anesthesia induction until extubation
Measure: Median (Inter-Quartile Range); unit: micrograms
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 49 | 47
micrograms | 350 [250 to 418.8] | 350 [300 to 450]

ADVERSE EVENTS:
Time Frame: During the hospital length of stay up to one week.
Groups:
- Desflurane: Patients will receive desflurane as general anesthetic
  propofol or desflurane: comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
- Propofol: Patients will receive propofol as general anesthetic
  propofol or desflurane: comparison of the incidence in delirium and post-operative cognitive dysfunction from propofol and desflurane in patients under general anesthesia
Arm/Group | Desflurane | Propofol
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No